CLINICAL TRIAL: NCT00753649
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Infanrix Hexa Vaccine in Healthy Infants
Brief Title: Immunogenicity and Safety of GSK Biologicals' Infanrix Hexa in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103506; 2013-003428-34 (EudraCT Number)
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis B; Tetanus; Poliomyelitis; Diphtheria; Haemophilus Influenzae Type b; Acellular Pertussis
Keywords: Infant; First nation; Aboriginal; Canada
MeSH Terms: conditions — Hepatitis B; Tetanus; Poliomyelitis; Diphtheria; Haemophilus Infections

ARMS (2):
- Aboriginal infants group (Experimental)
  Interventions: Biological: Infanrix™ hexa
- Other Non-Aboriginal infants (Active Comparator)
  Interventions: Biological: Infanrix™ hexa

INTERVENTIONS:
Biological: Infanrix™ hexa — Intramuscular, three doses
  Other Names: DTPa-HBV-IPV/Hib

SUMMARY:
This study will evaluate GSK Biologicals' DTPa-HBV-IPV/Hib vaccine given as a three-dose primary vaccination course at 2, 4 and 6 months of age, in terms of safety and immunogenicity in different population of infants residing in Canada.

DETAILED DESCRIPTION:
This protocol posting has been updated following Protocol amendment 1 (19-MAY-2010).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent/guardian can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Healthy subjects as established by medical history before entering into the study.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs from birth until first primary vaccination dose..
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Major congenital defects or serious chronic illness.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B and/or Hib vaccination or disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* The following condition is temporary or self limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:
* Current febrile illness or axillary temperature of ≥ 37.5 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2008-09-23 (Actual); Primary Completion 2013-03-12 (Actual); Study Completion 2013-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=19621

REFERENCES:
- [Background] Scheifele DW, Ferguson M, Predy G, Dawar M, Assudani D, Kuriyakose S, Van Der Meeren O, Han HH. Immunogenicity and safety of 3-dose primary vaccination with combined DTPa-HBV-IPV/Hib vaccine in Canadian Aboriginal and non-Aboriginal infants. Vaccine. 2015 Apr 15;33(16):1897-900. doi: 10.1016/j.vaccine.2015.02.015. Epub 2015 Feb 18. PMID 25701314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started on 23-Sep-2008 and enrolled 224 subjects from Canada.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix Hexa Aboriginal Group: Subjects of aboriginal origins who received 3 doses of Infanrix Hexa vaccine at 2, 4, and 6 months of age, administered as an intramuscular injection into the right side of the thigh. Subjects also received two doses of Rotarix vaccine at 2 and 4 months of age (administered orally), a pneumococcal conjugate vaccine, meningococcal serogroup C conjugate vaccine and an influenza vaccine according to the recommended provincial infant immunisation schedules.
- Infanrix Hexa Non-Aboriginal Group: Subjects of non-aboriginal origins who received 3 doses of Infanrix Hexa vaccine at 2, 4, and 6 months of age, administered as an intramuscular injection into the right side of the thigh. Subjects also received two doses of Rotarix vaccine at 2 and 4 months of age (administered orally), a pneumococcal conjugate vaccine, meningococcal serogroup C conjugate vaccine and an influenza vaccine according to the recommended provincial infant immunisation schedules.
Period: Overall Study
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Started | 112 | 112
Completed | 105 | 112
Not Completed | 7 | 0
Not completed — Migrated/moved from study area | 1 | 0
Not completed — Lost to follow-up-incomplete vaccination | 3 | 0
Not completed — Lost to follow-up-complete vaccination | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.3 (1.38) | 9.2 (1.3) | 9.25 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 52 | 114
  Male | 50 | 60 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol Phosphate (Anti-PRP)
Description: A seroprotected subject was a subject whose anti-PRP antibody concentration was greater or equal to (≥) 0.15 microgram per milliliter (µg/mL).
Time Frame: One month after (POST) Dose 3.
Population: The analysis was performed on the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received 3 doses of Infanrix Hexa vaccine and for whom data concerning immunogenicity outcome measures were available.
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 94 | 107
Subjects | 92 | 106

2. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥1µg/mL
Description: For this assay, 1 μg/mL was considered as the seropositivity cut-off.
Time Frame: One month after (POST) Dose 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 94 | 107
Subjects | 83 | 91

3. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Anti-PRP antibody concentrations were presented as Geometric mean Concentrations (GMC), expressed as micrograms per milliliter (μg/mL).
Time Frame: One month after (POST) Dose 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 94 | 107
µg/mL | 6.123 [4.498 to 8.334] | 3.51 [2.745 to 4.488]

4. Secondary Outcome: Number of Seroprotected Subjects Against Hepatitis B (Anti-HBs)
Description: A seroprotected subject was a subject with anti-HBs antibody concentrations ≥ 10 milli-International Units ler milliliter (mIU/mL). A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis. Some of the available blood samples initially tested with ELISA were re-tested using the new assay, CLIA.
Time Frame: One month after (POST) Dose 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 91 | 103
Subjects | 91 | 103

5. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations ≥100 mIU/mL
Description: The testing was done using the Enzyme-Linked Immunosorbent assay (ELISA) assay.
Time Frame: One month after (POST) Dose 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 91 | 103
Subjects | 89 | 100

6. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Anti-HBs antibody concentrations were assessed by Enzyme-Linked Immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs).
Time Frame: One month after (POST) Dose 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 91 | 103
mIU/mL | 1797.9 [1375.1 to 2350.7] | 1544.4 [1210.4 to 1970.5]

7. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31 day (Days 0-30) post vaccination
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with at least one dose of Infanrix hexa administration documented.
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 112 | 112
Subjects | 26 | 19

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period up to Last subject last visit on 03/12/2013
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Number analyzed (Participants) | 112 | 112
Subjects | 6 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs during the 31-day post-vaccination period, SAEs during the entire period up to Last subject last visit on 03/12/2013.
Description: During this study, no solicited adverse events were collected, therefore none are reported.
Arm/Group | Infanrix Hexa Aboriginal Group | Infanrix Hexa Non-Aboriginal Group
Serious Adverse Events (participants affected / at risk) | 6/112 | 0/112
Other Adverse Events (participants affected / at risk) | 6/112 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa Aboriginal Group (N=112) | Infanrix Hexa Non-Aboriginal Group (N=112)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa Aboriginal Group (N=112) | Infanrix Hexa Non-Aboriginal Group (N=112)
Pyrexia (General disorders) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.